CLINICAL TRIAL: NCT05676203
Title: A Randomised, Phase 3 Trial Comparing 3-weekly Docetaxel 75 mg/m2 (in a 3 Week Cycle) Versus 2-weekly Docetaxel 50 mg/m2 (in a 4 Week Cycle) in Combination With Darolutamide + ADT in Patients With mHSPC
Brief Title: A Trial Comparing Docetaxel 75 mg/m2 (3w) Versus Docetaxel 50 mg/m2 (2w) in Combination With Darolutamide + ADT in mHSPC Patients
Acronym: ARASAFE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jena University Hospital (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Marc-Oliver Grimm, Prof. Dr. Marc-Oliver Grimm, Jena University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UTN-01-2022
Record Dates: First submitted 2022-12-14; First posted 2023-01-09 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Hormone-Sensitive Prostate Cancer (mHSPC)
Keywords: prostate cancer; metastatic prostate cancer; metastatic hormone-sensitive prostate cancer; docetaxel; darolutamide; safety
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Active Comparator): 6 x Docetaxel 75 mg/m2 every 3 weeks of a 3 week cycle Co-administration of docetaxel, darolutamide and standard ADT
  Interventions: Drug: Standard ADT (androgen deprivation therapy); Drug: Standard Darolutamide; Drug: Docetaxel
- Arm 2 (Experimental): 6 x Docetaxel 50 mg/ m2 every 2 weeks of a 4 week cycle Co-administration of docetaxel, darolutamide and standard ADT
  Interventions: Drug: Standard ADT (androgen deprivation therapy); Drug: Standard Darolutamide; Drug: Docetaxel

INTERVENTIONS:
Drug: Standard ADT (androgen deprivation therapy) — as prescribed by the treating physician.
Drug: Standard Darolutamide — 2x600 mg/d as prescribed by the treating physician
Drug: Docetaxel — Docetaxel

SUMMARY:
The purpose of this clinical phase 3 randomized trial is to compare two different dosing schedules of Docetaxel in combination with ADT and Darolutamide in subjects with mHSPC. The main question aims to compare grade 3-5 adverse events (AEs) in patients with mHSPC treated with 6 cycles of either Docetaxel 75 mg/m2 every 3 weeks in a 3 week cycle or 6 cycles of Docetaxel 50 mg/m2 every 2 weeks in a 4 week cycle in combination with Darolutamide + ADT. The primary endpoint are Grade 3-5 AEs, followed by neutropenia grade 3/4 + grade 5 AEs to be analysed 28 weeks after last patient first Docetaxel dose (LPFD).

DETAILED DESCRIPTION:
This is a randomized, open, controlled, multicenter phase III clinical trial. Approximately 250 patients with mHSPC who are candidates for docetaxel, darolutamide and ADT will be randomized (1:1 ratio) to one of the following study arms:

* Arm 1: 6 x Docetaxel 75 mg/m2 every 3 weeks of a 3 week cycle
* Arm 2: 6 x Docetaxel 50 mg/ m2 every 2 weeks of a 4 week cycle Subjects will be stratified at randomization for the extent of disease and for Alkaline Phosphatase levels.

All subjects must receive ADT of Investigator's choice (LHRH agonist/antagonists or orchiectomy) and darolutamide as standard therapy. Six cycles of docetaxel are be administered after randomization according to either Arm 1 or Arm 2. After completion of study drug treatment, subjects will continue with the observation period. During the observation period all subjects will continue with Darolutamide+ADT until occurrence of metastatic castration-resistant prostate cancer (mCRPC).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Males ≥18 years of age
* Histologically or cytologically confirmed adenocarcinoma of prostate
* Investigator assessed metastatic disease documented either by a positive bone scan, or for soft tissue or visceral metastases, either by contrast-enhanced abdominal/pelvic/chest computed tomography (CT) or magnetic resonance imaging (MRI) scan assessed. Metastatic disease is defined as either malignant lesions in bone scan or soft tissue/visceral lesions according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1. Lymph nodes are measurable if the short axis diameter is ≥15 mm, soft tissue/visceral lesions are measurable if the long axis diameter is ≥10 mm.
* Subjects with lymph node metastases only (either below the aortic bifurcation (N1) or above the aortic bifurcation (M1a)) will not be eligible for the study.
* Subjects must be candidates for ADT, docetaxel and darolutamide therapy per Investigator's judgment
* Started ADT (LHRH agonist/antagonist or orchiectomy) with or without first generation anti-androgen, but no longer than 12 weeks before randomization. For subjects receiving LHRH agonists, treatment in combination with a first generation anti-androgen for at least 4 weeks, prior to randomization is recommended. First generation anti-androgen has to be stopped prior to randomization.
* An Eastern Cooperative Oncology Group performance status of 0 or 1
* Blood counts at Screening: hemoglobin ≥9.0 g/dL, absolute neutrophil count ≥1.5x109/L, platelet count ≥100x109/L (subject must not have received any growth factor within 4 weeks or a blood transfusion within 7 days of the hematology laboratory sample obtained at Screening)
* Screening values of serum alanine aminotransferase and/or aspartate transaminase ≤1.5x upper limit of normal (ULN), total bilirubin ≤ULN, creatinine ≤2.0x ULN

Sexually active male subjects must agree to use condoms as an effective barrier method and refrain from sperm donation, and/or their female partners of reproductive potential to use a method of effective birth control, during the treatment with darolutamide and for 3 months after the end of the treatment with darolutamide and 6 months after treatment with docetaxel.

Exclusion Criteria:

* Exclusion criteria
* Prior treatment with:
* LHRH agonist/antagonists started more than 12 weeks before randomization Second-generation androgen receptor (AR) inhibitors such as enzalutamide, apalutamide, darolutamide, other investigational AR inhibitors
* Cytochrome P 17 enzyme inhibitor such as abiraterone acetate or oral ketoconazole as antineoplastic treatment for prostate cancer
* Chemotherapy, immunotherapy, radium or other therapeutic radiopharmaceuticals for prostate cancer (e.g. Lutetium177-PSMA) prior to randomization
* Treatment with radiotherapy (external beam radiation therapy, brachytherapy) within 2 weeks before randomization
* Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation of the study drugs
* Contraindication to both CT and MRI contrast agent
* Had any of the following within 6 months before randomization: stroke, myocardial infarction, severe/unstable angina pectoris,coronary/peripheral artery bypass graft, congestive heart failure (New York Heart Association Class III or IV)
* Uncontrolled hypertension as indicated by a resting systolic blood pressure (BP) ≥160 mmHg or diastolic BP ≥100 mmHg despite medical management
* Had a prior malignancy. Adequately treated basal cell or squamous cell carcinoma of skin or superficial bladder cancer that has not spread behind the connective tissue layer (i.e., pTis, pTa, and pT1) is allowed, as well as any other cancer for which treatment has been completed ≥5 years before randomization and from which the subject has been disease-free
* A gastrointestinal disorder or procedure which is expected to interfere significantly with absorption of study drug
* An active viral hepatitis, known human immunodeficiency virus infection with detectable viral load, or chronic liver disease with a need for treatment
* Previous (within 28 days before the start of study drug or 5 half-lives of the investigational treatment of the previous study, whichever is longer) or concomitant participation in another clinical study with investigational medicinal product(s)
* Any other serious or unstable illness, or medical, social, or psychological condition, that could jeopardize the safety of the subject and/or his/her compliance with study procedures, or may interfere with the subject's participation in the study or evaluation of the study results
* Inability to swallow oral medications
* Previous assignment to treatment in this study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Rate of grade 3-5 AEs | 28 weeks after last patient first Docetaxel dose (LPFD)
  Rate of grade 3-5 AEs, followed by rate of neutropenia grade 3/4 + grade 5 AEs t

SECONDARY OUTCOMES:
PSA-response | 28 after LPFD
  PSA-response (PSA <=0.2, >0.2-4.0 und >4.0 ng/ml) determined at week 28 after LPFD
Time to castration-resistant prostate cancer | approximately 42 months
  approx. every 90 days, defined as the time to PSA progression with serum testosterone being at castrate level <0.50 ng/mL, or the time to progression by soft tissue/visceral lesions or time to progression by bone lesions whatever comes first;
Overall survival | approximately 42 months
  defined as the time (in days) from date of randomization until death from any cause
Time to initiation of subsequent antineoplastic therapy | approximately 42 months
  approx. every 90 days up to the date of first subsequent antineoplastic therapy for prostate cancer
Symptomatic skeletal event free survival (SSE) | approximately 42 months
  approx. every 90 days up to the first occurence of SSE, symptomatic skeletal event free survival, defined as the time from randomization to the first occurrence of SSE or death from any cause, whichever comes first. An SSE is defined as EBRT to relieve skeletal symptoms, or new symptomatic pathologic bone fracture, or occurrence of spinal cord compression or tumor-related orthopedic surgical intervention, whichever comes first.
Time to first symptomatic skeletal event (SSE) | approximately 42 months
  approx. every 90 days up to the first occurence of SSE, defined as the time from randomization to the first occurrence of SSE. An SSE is defined as EBRT to relieve skeletal symptoms, or new symptomatic pathologic bone fracture, or occurrence of spinal cord compression or tumor-related orthopedic surgical intervention, whichever comes first.
Time to pain progression | approximately 42 months
  approx. every 90 days up to the first date a subject experiences a pain progression. Pain to be assessed with a patient reported questionaire
Time to worsening of physical symptoms of disease | approximately 42 months
  approx. every 90 days up to the first date a subject experiences an increase in physical symptoms based on the NCCN-FACT-FPSI-17 questionnaire
Treatment emergent adverse events | approximately 42 months
  all grade AEs until the end-of-study treatment visit (to be analysed 26 weeks after last patient first Docetaxel, all grade AEs until the discontinuation visit, all and Study drug-related SAEs until the end of Survival Follow-up

CONTACTS AND LOCATIONS:
Locations (43):
- Austria (2):
  - Ordensklinikum Linz GmbH, Elisabethinen, Linz
  - Krankenhaus der Barmherzigen Brüder, Vienna
- Germany (41):
  - Nationales Centrum für Tumorerkrankungen (NCT) Heidelberg, Heidelberg, Baden-Wurttemberg
  - Klinikum Wetzlar, Wetzlar, Hesse
  - Med. Hochschule Hannover, Hanover, Lower Saxony
  - Urologische Klinik München Planegg, Planegg, München
  - Urologicum Duisburg, Duisburg, North Rhine-Westphalia
  - Brüderkrankenhaus St- Josef Paderborn, Paderborn, North Rhine-Westphalia
  - Urologisches Zentrum Euregio, Würselen, North Rhine-Westphalia
  - Krankenhaus Martha-Maria Halle Dölau gGmbH, Halle, Saxony-Anhalt
  - Praxisgemeinschaft f. Onkologie & Urologie, Wilhelmshaven, Schleswig-Holstein
  - University Hospital Jena, Department of Urology, Jena, Thuringia
  - Marien Krankenhaus, Bergisch Gladbach
  - Vivantes Prostatazentrum im Klinikum am Urban, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Urologie Schlosscarree, Braunschweig
  - UROLOGIE BAYENTHAL Gemeinschaftspraxis, Cologne
  - Städtisches Klinikum Dessau, Dessau
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Helios Klinikum Erfurt, Erfurt
  - Uniklinikum Erlangen, Erlangen
  - KEM | Evang. Kliniken Essen-Mitte, Essen
  - Universitätsklinikum Essen, Essen
  - Krankenhaus Nordwest, Frankfurt am Main
  - Universitäts Klinikum Frankfurt, Frankfurt am Main
  - Universitätsklinikum Giessen und Marburg GmbH, Standort Giessen, Giessen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - St. Anna Hospital Herne, Herne
  - Universitätsklinikum Schleswig-Holstein - Campus Lübeck, Lübeck
  - Universitätsklinikum Magdeburg, Magdeburg
  - Universitätsmedizin Mannheim, Mannheim
  - Universitätsklinikum Gießen und Marburg - Standort Marburg, Marburg
  - LMU Klinikum, München
  - TUM Klinikum, München
  - Universitätsklinikum Münster, Münster
  - Klinikum Nürnberg, Nuremberg
  - St. Theresien Krankenhaus Nürnberg, Nuremberg
  - Studienpraxis Urologie, Nürtingen
  - Brüderkrankenhaus, Trier
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - Helios Universitätsklinikum Wuppertal, Wuppertal
  - Uniklinikum Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No